| Pharmacokinetic Modeling of Ropivacaine Following Single Shot Erector Spinae Pla | ne |
|---|---|
| Block in Anesthetized Children | |

**NCT:** 04298099

Date: 2/17/2021 (date of original analysis document)

## **Statistical Analysis:**

Prior investigations have suggested that a 1-compartment model with an absorption rate constant best describes the pharmacokinetic profile of Ropivacaine. Therefore, population pharmacokinetic analysis was performed with NONMEM v.7.4<sup>12,13</sup> (Icon, PLC; Dublin, Ireland) and PDx-Pop 5.2 (Icon, PLC, Dublin, Ireland) using first-order conditional estimation with interaction (FOCE-I). One- and two-compartment models with an absorption rate constant (Ka<sup>-1</sup>) and various error structures were evaluated, and the final model was selected based upon a significant reduction in the objective function value (p<0.05), in conjunction with standard subjective evaluation of graphical representations of model fit. Models were generated for both total and free Ropivacaine concentrations. After the final models were generated, simulation (n=1000) of serum concentrations (total and free Ropivacaine) was performed using 1, 1.5, 2, and 2.5 mg/kg/dose in a patient with a median weight value from the dataset.

## **REFERENCES:**

- 1. Richebé P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. *Anesthesiology*. 2018; 129(3):590-607.
- 2. Lönnqvist PA, Ecoffey C, Bosenberg A, et al. The European society of regional anesthesia and pain therapy and the American society of regional anesthesia and pain medicine joint committee practice advisory on controversial topics in pediatric regional anesthesia I and II: what do they tell us? *Curr Opin Anaesthesiol*. 2017; 30(5):613-620.

- 3. Taenzer AH, Herrick M, Hoyt M, et al. Variation in pediatric local anesthetic dosing for peripheral nerve blocks: an analysis from the Pediatric Regional Anesthesia Network (PRAN). *Reg Anesth Pain Med.* 2020; 45(12):964-969.
- 4. Suresh S, De Oliveira GS Jr. Local anaesthetic dosage of peripheral nerve blocks in children: analysis of 40 121 blocks from the Pediatric Regional Anesthesia Network database. *Br J Anaesth*. 2018; 120(2):317-322.
- 5. L Long JB, Birmingham PK, De Oliveira GS Jr, et al. Transversus abdominis plane block in children: a multicenter safety analysis of 1994 cases from the PRAN (Pediatric Regional Anesthesia Network) database. *Anesth Analg.* 2014; 119(2):395-9.
- 6. Knudsen K, Beckman Suurküla M, Blomberg S, et al. Central nervous and cardiovascular effects of i.v. infusions of Ropivacaine, bupivacaine and placebo in volunteers. *Br J Anaesth*. 1997; 78(5):507-14.
- 7. Forero M, Adhikary SD, Lopez H, et al. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. *Reg Anesth Pain Med*. 2016; 41(5):621-7.
- Suresh S, De Oliveira GS Jr. Blood Bupivacaine Concentrations After Transversus Abdominis
  Plane Block in Neonates: A Prospective Observational Study. *Anesth Analg.* 2016; 122(3):814-7.
- 9. Yasumura R, Kobayashi Y, Ochiai R. A comparison of plasma levobupivacaine concentrations following transversus abdominis plane block and rectus sheath block. *Anaesthesia*. 2016; 71(5):544-9.
- Berde CB, Yaster M, Meretoja O, et al. Stable plasma concentrations of unbound Ropivacaine during postoperative epidural infusion for 24-72 hours in children. *Eur J Anaesthesiol*. 2008; 25(5):410-7.

- 11. Arvidsson T, Eklund E. Determination of free concentration of Ropivacaine and bupivacaine in blood plasma by ultrafiltration and coupled-column liquid chromatography. *J Chromatogr B Biomed Appl.* 1995; 668(1):91-8.
- 12. Ollier E, Heritier F, Bonnet C, et al. Population pharmacokinetic model of free and total Ropivacaine after transversus abdominis plane nerve block in patients undergoing liver resection. *Br J Clin Pharmacol*. 2015; 80(1):67-74.
- 13. Walker BJ, Long JB, Sathyamoorthy M, et al. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. *Anesthesiology*. 2018; 129(4):721-732.
- 14. Aarons L, Sadler B, Pitsiu M, et al. Population pharmacokinetic analysis of Ropivacaine and its metabolite 2',6'-pipecoloxylidide from pooled data in neonates, infants, and children. Br J Anaesth. 2011; 107(3):409-24.
- 15. Bo"senberg AT, Thomas J, Cronje L, et al. Pharmacokinetics and efficacy of Ropivacaine for continuous epidural infusion in neonates and infants. *Paediatr Anaesth*. 2005; 15: 739–49.